CLINICAL TRIAL: NCT02777853
Title: Can Tea Prevent Impairments in Vascular Function and Insulin Sensitivity Induced by 7-days Physical Inactivity and Overfeeding in Healthy Men
Brief Title: The Effect of Tea on Vascular Function and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, Kirsty Woodward, PhD Student, Liverpool John Moores University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Greenshield16
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Insulin Resistance
Keywords: tea; cardiovascular; vascular; metabolism; microcirculation; physical inactivity; polyphenols; conduit artery; endothelial function; cerebrovascular; insulin sensitivity
MeSH Terms: conditions — Insulin Resistance; Sedentary Behavior | interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (green) tea (Experimental): Tea to be ingested 3 times per day for 7 days.
  Interventions: Dietary Supplement: Green tea
- Placebo tea (Placebo Comparator): Tea to be ingested 3 times per day for 7 days.
  Interventions: Dietary Supplement: Placebo tea

INTERVENTIONS:
Dietary Supplement: Green tea — The intervention product is regular green tea brewed with hot water in a large quantity. The tea obtained is dried and the powder, with added sugar, is distributed over sealed aluminium sachets (1 gram of powder per sachet). The product has been cleared for consumption by Unilever's Microbiology Department and the independent Safety and Environmental Assurance Centre of Unilever.
  Other Names: Camillia sinesis
  Arms: Active (green) tea
Dietary Supplement: Placebo tea — A product of similar colour and taste, but not the presumed actives of tea (polyphenols), is used as placebo. The product has been cleared for consumption by Unilever's Microbiology Department and the independent Safety and Environmental Assurance Centre of Unilever.
  Arms: Placebo tea

SUMMARY:
The aim of this research is to explore changes in peripheral/cerebrovascular function and insulin sensitivity after a 7-day combination of physical activity reduction (-50% steps per day) and overfeeding (+50% kcal per day, comprising 65% fat) in healthy male volunteers, and examine whether daily intake of tea can prevent such changes.

DETAILED DESCRIPTION:
The aim of this study is to explore the impact of a 7-day 'unhealthy' lifestyle that combines physical activity reduction (-50% steps per day) and overfeeding (+50% kcal per day, comprising 65% fat) on peripheral (conduit artery and skin microvessels) and cerebrovascular function and insulin sensitivity in healthy male participants. Moreover, the investigators will explore whether the detrimental impact of this lifestyle can be mitigated by daily tea consumption (equivalent to 6 cups/day). To explore this hypothesis, the investigators will perform measurements of these parameters before and after 7-days of reduced physical activity and overfeeding, with and without the combination of daily tea ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years
* Male
* Habitually active (>8,000 steps/day)
* Healthy

Exclusion Criteria:

* Smokers
* Medical history of cardiovascular/metabolic disease
* Family history of cardiovascular disease (first degree relatives)
* On medication known to influence the cardiovascular system
* BMI of <18 or >30 kg/m2
* Known food allergies or special dietary requirements
* Vaccination (<1 week) due to induced systemic inflammatory reaction

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Post 7 day intervention
  This will be measured following a carbohydrate-rich meal tolerance test (MTT) after an overnight fast, combined with regular venous blood sampling of insulin and glucose.

SECONDARY OUTCOMES:
Vascular function | Post 7 day intervention
  Peripheral vascular function will be measured via endothelial-dependent flow-mediated dilation (FMD) of the brachial and femoral arteries, with microcirculatory function being assessed using local thermal hyperaemia and laser Doppler flowmetry (LDF), in addition to full-field laser perfusion imaging (FLPI). Cerebrovascular function will be examined via transcranial Doppler.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty A Woodward, BSc, Principal Investigator — Liverpool John Moores University
Locations (1):
- Research Institute for Sport and Exercise Sciences (RISES), Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No